CLINICAL TRIAL: NCT01598714
Title: A Comparison of Patient Satisfaction Between Darco, Podalux and Standard Dressing Shoes Following Forefoot Surgery
Brief Title: Comparison of Patient Satisfaction Between 3 Types Dressing Shoes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH15909
Record Dates: First submitted 2012-05-03; First posted 2012-05-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Patients Requiring Forefoot Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Darco shoe (Other): Darco walking shoe provided
  Interventions: Device: Darco shoe
- Podalux Shoe (Other): Podalus shoe
  Interventions: Device: Podalux shoe
- Standard dressing shoe (Other): Standard dressing shoe
  Interventions: Device: Standard dressing shoe

INTERVENTIONS:
Device: Darco shoe — Darco shoe
  Arms: Darco shoe
Device: Podalux shoe — Podalux shoe
  Arms: Podalux Shoe
Device: Standard dressing shoe — Standard dressing shoe
  Arms: Standard dressing shoe

SUMMARY:
This study compares patient satisfaction in terms of pain relief, mobility and ease of use between 3 commonly used types of post-surgical footwear. This study randomises patients who participate into one of 3 groups of footwear, namely Darco, Podalux or standard dressing shoe. Number of patients enrolled is determined by power calculation. Patients complete a single, simple previously validated questionnaire the MOXFQ (Manchester-Oxford Foot Questionnaire) at their 6 week follow-up appointment and statistical differences between the group are calculated using a significance level of p<0.05. This study will help us determine the best foot-wear to offer the investigators post-surgical patients.

This study will form original research.

DETAILED DESCRIPTION:
Methodology:

This will be a randomised trial with three arms: 1. Darco, 2. Podalux, 3. Standard dressing shoe.

Design:

A randomised controlled trial will ensure that shoes are distributed without surgeon bias, and will be performed prior to surgery by the principle investigator. Baseline differences will be assessed for by administration of a pre-operative MOXFQ score prior to randomisation. Primary outcome measure will be difference in score between groups post-operatively, however we will also analyse the absolute change in score between groups, although this we do not feel can be the primary outcome measure as the major reason for the change in MOXFQ from pre to post operation will be the surgery itself.

Blinding and randomisation:

Randomisation will be achieved by a computer generated randomisation table. As two main types of surgery will be used in the study as outlined below (namely 1st metatarsal osteotomy and 1st MTP joint fusion), we will have two separate randomisation groups to ensure that numbers of each operation are evenly distributed between the three types of shoe. This will improve heterogeneity of the groups. We have decided to use two types of surgery as the research question is relevant to both and we can perform a secondary analysis to look between these groups more closely as detailed below. For practical purposes this will not be a blinded trial as the surgeon and patient will both be aware of the shoe provided.

Analysis:

We have sought an opinion from a statistician. The data for the MOXFQ (primary outcome measure) will be subdivided into the 3 domains, walking/standing, pain and social demain, and the raw scores will be treated as laid out in the original paper by Dawson et al. (2011) [2].

The scores from each of the 3 domains is then converted to a metric 0-100 scale for analysis.

The Surgical Show Questionnaire scores (secondary outcome measure) will be totalled to give a score out of 50.

The data will be analysed for normality, and comparison will be made using the ANOVA or Kruskall-Wallis testing for unpaired continuous data as advised by the statistician, with a significance level set at P<0.05.

We have been advised that we can perform a secondary analysis using linear regression to look at the effect of the differences within the groups on outcome, for example differences between operation type and each of the shoes.

Statsdirect statistical software will be used. There is a question (Q1) in the Surgical Shoe Questionnaire that asks the patient how long they wore the shoe for. This question is not included in the scoring and is included to assess for patient use, and will be used as a secondary outcome measure. The study does not necessarily require strict patient compliance as discontinuation of the shoe is valuable information in its own right. This can be looked at within the secondary analysis using linear regression as well.

The primary analysis will be intention to treat analysis.

Outcome Measures:

The MOXFQ is a widely validated foot score used in the assessment of the foot with 3 specified domains; walking/standing, pain, and social interaction (Appendix 1). The MOXFQ (Manchester-Oxford foot Questionnaire) walking/standing domain will be used as the primary outcome measure as this includes the questions that are most relevant to ease of shoe use. However the other 2 domains will be analyses although there is more likely to be confounding factors that will affect these. Secondary outcome measures will include 11 questions related to the wearing of the shoe forming a separate questionnaire. (Appendix 2).

Setting:

The setting for the study will be clinical. Out-patients clinic for recruitment and follow-up and theatre for randomisation and post-surgical shoe provision.

Participants:

Patients will be recruited from outpatient clinics directly by the clinical care team, and will be recruited from those who have been listed for forefoot surgery.

Patients undergoing forefoot surgery who meet the inclusion criteria will be invited to participate in the trial and provided with written information within the clinic setting [see Patient Information Sheet ver 1.0]. Those wishing to participate will be asked to provide written consent on the day of surgery [see Patient Consent Form ver 1.0] which will be undertaken by the principle investigator.

Inclusion and exclusion criteria have been chosen that include the majority of patients undergoing straightforward forefoot surgery who would be normally managed in our current post-operative shoe (the Darco), and who have capacity to consent to surgery.

Inclusions:

Patients over 18 years age Patients normally independently mobile Patients with no significant co-morbidities that would be expected to affect normal ambulation Patients undergoing straightforward 1st ray surgery eg. 1st MTPJ arthrodesis, 1st metatarsal osteotomy, (in combination with 2nd ray procedures allowed) Patients able to understand and complete questionnaires

Exclusions:

Patients under 18 years age Patients not independently mobile Patients with significant co-morbidities that effect normal ambulation (eg hip arthritis) Patients undergoing complicated forefoot reconstructive surgery or surgery on rays other then 1st and 2nd.

Patients unable to understand or complete self-administered questionnaires

Sampling:

Sample size will be determined based on a power calculation using MOXFQ (Manchester-Oxford foot Questionnaire) as the primary outcome measure. The MOXFQ is a widely validated foot score used in the assessment of the foot with 3 specified domains; walking/standing, pain, and social interaction (Appendix 1). It is the walking/standing domain that has provided us with the data for the power calculation (1,2).

The walking/standing domain scores out of 35 which is then transformed to a score out of 100, an approximate multiple of 3.

We have calculated the standardised difference as 15 out of 100, which equates to a raw score of 30 out of 35, or a one point drop for 5 out of 7 questions, which is the minimum difference we wish to detect.

Using a significance level of 0.05 and power level of 0.8 we calculate each arm of the trial will consist of 29 patients (standardised difference between means =15, standard deviation =20). This has been agreed with the statistician.

In total 90 patients will be required. We estimate approximately 6 to 8 of these procedures are carried out with the Foot and ankle unit per week, and therefore estimate the study will take around 12 to 16 weeks to complete.

Subject with-drawl:

Subjects are free to with-draw at any time during the study, and will be included in the intention to treat analysis by being assigned a questionnaire score identical to that of the lowest scoring participant in their randomisation group. For example if the Darco group score from 65 to 95 of the MOXFQ, a subject who withdraws will be assigned a value of 65. Due to the short nature of the study we anticipate this will be infrequent. Those patients who change their surgical footwear will be included in the intention to treat analysis for their original randomised group as agreed with the statistician.

Intervention:

Once patients have consented and completed the pre-operative MOXFQ score, following their surgery, patients will be randomly assigned to one of the three treatment arms to wear the shoe for 6 weeks following their surgery. The participant will be advised that withdrawal from the study at any stage is possible and only data collected up until that point will be used, although due to the timeframe and nature of the study we believe this is unlikely to occur.

Patients will attend for their routine follow-up at 2 weeks post-surgery for wound review and removal of any sutures used in our nurse-led dressing clinic.

Patients will attend for their routine 6 week post-surgery follow-up appointment with their consultant and will be asked to complete the questionnaire assessment. This will mark the end of the study.

Safety assessments:

Whilst we do not anticipate any adverse events, any problems with the shoes will be monitored during the clinic visits and documented for the study.

Quality control:

The study will be overseen by the principle investigator. All questionnaires will be looked at as soon as they are completed in clinic, to ensure completeness.

Project management The study is straightforward, with minimum man-power requirements, and will therefore be conducted by the principle and co-investigators. Progress will be monitored at the regular meetings of the foot and ankle research group held every 2 months. Data will be held within the secured office of the foot and ankle fellow, and be stored anonymously using a participant number assigned on consent. The master patient log with the participants details will be held as a paper copy within the foot and ankle office.

Expertise As this study only involves the administration of a simple questionnaire, no specialist involvement is required.

Ethical Issues The patient information leaflet is provided to patients when they are listed for surgery in clinic to allow them time to consider participating in the trial. Patients happy to participate in the trial are consented on the day of surgery by the lead or co-investigators. Patients are allocated a particpant number held on a master log in a locked office, and throughout the trial questionnaires use this number to maintain confidentiality as per Caldicott guidelines.

Costing Schedule No additional costs will be incurred. The Darco and standard dressing shoes are already in use in the hospital, and the Podalux shoes have been provided on a free trial basis by Donjoy Int. Basic costs such as photocopying questionnaires will be provided by the foot and ankle research unit.

Funding arrangements The only additional funding we anticipate is with the provision of questionnaires and is estimated at around £36.00 (based on the price of photocopying 5p per sheet). This includes 90 consent forms (1 page), 90 (4 pages), 180 MOXFQ's (1 page), 90 Surgical shoe questionnaires (1page).

We anticipate the role of the research nurse to be negligible as all the questionnaires and paperwork will be administed in the out-patients clinics or prior to surgery by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years age
* Patients normally independently mobile
* Patients with no significant co-morbidities that would be expected to affect normal ambulation
* Patients undergoing straightforward 1st ray surgery eg. 1st MTPJ arthrodesis, 1st metatarsal osteotomy, (in combination with 2nd ray procedures allowed)
* Patients able to understand and complete questionnaires

Exclusion Criteria:

* Patients under 18 years age
* Patients not independently mobile
* Patients with significant co-morbidities that effect normal ambulation (eg hip arthritis)
* Patients undergoing complicated forefoot reconstructive surgery or surgery on rays other then 1st and 2nd.
* Patients unable to understand or complete self-administered questionnaires

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (Outcome measure looking at foot pain,and function) | Change from baseline at 6 weeks post-operative
  Differences between the 2 groups in change from baseline in questionnaire score at 6 weeks post operative

SECONDARY OUTCOMES:
Surgical Shoe Questionnaire | 6 weeks post-operative
  Questionnaire designed with questions regarding confort, and ease of use of post-operative surgical shoes

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Davies, MBChB, Study Director — Sheffield Teaching Hospitals NHS Foundation Trust; Chris M Blundell, MBChB, Principal Investigator — Sheffield Teaching Hosiptals NHS Trust
Locations (1):
- Northern General Hospital, Sheffield, S Yorks, United Kingdom